CLINICAL TRIAL: NCT03893175
Title: Towards Predicting the Analgesic Response to Ibuprofen Following Third-molar Extraction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 832417
Record Dates: First submitted 2019-03-22; First posted 2019-03-28 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Impacted Third Molar Tooth; Pain, Acute
Keywords: Non-steroidal anti-inflammatory drugs
MeSH Terms: conditions — Acute Pain | interventions — Ibuprofen; Acetaminophen; Oxycodone

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either ibuprofen or placebo after third molar extraction when pain intensity is at least 4/10.
  Four hours after the masked ibuprofen or placebo, all subjects will receive open-label ibuprofen + acetaminophen to be taken every 4 hours for the first 2 days and then as needed for up to 7 days after oral surgery.
  Oxycodone will be available as a rescue medication if additional analgesic is requested.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Administration of ibuprofen vs. placebo will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen (Experimental): During the double-blind stage, subjects will receive blinded ibuprofen (400 mg by mouth) when pain is at least 4/10 following third molar extraction.
  During the open-label stage, all subjects will receive ibuprofen (400 mg by mouth) and acetaminophen (500 mg by mouth) to be taken every 4 hours around the clock for the first 2 days after third molar extraction and then as needed for pain up to 7 days after third molar extraction.
  Rescue medication (oxycodone 5 mg by mouth) will be available if additional analgesic is requested.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen; Drug: Oxycodone
- Placebo (Placebo Comparator): During the double-blind stage, subjects will receive blinded placebo when pain is at least 4/10 following third molar extraction.
  During the open-label stage, all subjects will receive ibuprofen (400 mg by mouth) and acetaminophen (500 mg by mouth) to be taken every 4 hours around the clock for the first 2 days after third molar extraction and then as needed for pain up to 7 days after third molar extraction.
  Rescue medication (oxycodone 5 mg by mouth) will be available if additional analgesic is requested.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen; Drug: Placebo; Drug: Oxycodone

INTERVENTIONS:
Drug: Ibuprofen — 400 mg by mouth every 4 hours for 2 days after third molar extraction and then as needed for pain up to 7 days after third molar extraction
  Other Names: Advil
Drug: Acetaminophen — 500 mg by mouth every 4 hours for 2 days after third molar extraction and then as needed for pain up to 7 days after third molar extraction
  Other Names: Tylenol
Drug: Placebo — By mouth
  Arms: Placebo
Drug: Oxycodone — 5 mg by mouth every 6 hours as needed for pain

SUMMARY:
This research study will evaluate inter-individual variability in the analgesic response to the non-steroidal anti-inflammatory drug (NSAID) ibuprofen after third molar extraction surgery. It will also investigate demographic, clinical, genetic, and environmental factors that cause this variability.

DETAILED DESCRIPTION:
The dramatic increase in opioid prescriptions over the past years has been linked to the concomitant rise in opioid addiction and to deaths from opioid abuse. Young adults' initial exposure to opioid analgesics is often following extraction of their impacted third molars, with an average of 5,000,000 cases in the USA per year. Over-prescribing of opioids for surgical pain, often 2-5 times more than patients actually use, further exacerbates this problem, as patients tend to save leftover pills rather than discard them. Up to 70% of individuals who become addicted to prescription opioids had access to leftover pills prescribed for others. This is particularly troubling as the odds of transitioning to heroin from prescription opioid abuse are much higher than other suspected gateway drugs, about 40 fold greater than non-gateway drug users. Heroin is now often laced with fentanyl derivatives making overdose and death more likely in even the most opioid tolerant individuals.

Multiple studies have demonstrated that non-addicting nonsteroidal anti-inflammatory drugs (NSAIDs) such as ibuprofen and diclofenac are effective in relieving pain after dental impaction surgery, being at least equally efficacious to optimal doses of immediate release opioid formulations combined with acetaminophen. However, these assessments of pain relief represent average scores and approximately 22% and 50% of individuals required additional opioid-containing rescue analgesics when ibuprofen and diclofenac were employed at FDA-approved dosages. A deeper understanding of the sources of variability in pain relief should allow improvements in the overall efficacy of NSAIDs by targeting treatment to those who are most likely to receive sufficient pain relief. Thus, optimizing pain therapy with NSAIDs by personalization would be expected to help limit the unnecessary prescription of highly addicting immediate release opioids. Moreover, these results may have applicability to other types of pain that are driven by inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women greater than 18 years of age requiring extraction of at least one impacted mandibular third molar tooth (at least 50% covered with bone).
* Body mass index (BMI) between 18 and 30 kg/m2.
* Absence of other major medical problems or contraindications to surgery or study drugs.
* Has not used tobacco products, including smoking cessation nicotine-containing products (e.g., nicotine patch, nicotine gum), for at least the 3 months prior to screening.
* Female subjects of child bearing potential must be using a medically acceptable method of contraception (oral contraception, Depo-Provera injection, IUD, condom with spermicide, diaphragm, cervical cap, progestin implant, abstinence, tubal ligation, oophorectomy, TAH) throughout the entire study period. All female subjects must consent to a urine pregnancy test at screening and a urine pregnancy test on the day of surgery, which must be negative at all time points.
* Has not ingested caffeine-containing products within 12 hours of surgery.
* All subjects must consent to a urine drug test at screening. Results must be negative. A positive result will be reported to the subject.
* Does not consume more than 1 alcoholic beverage per day on average.
* Subjects must reach a level of at least moderate pain within four hours of surgery completion, with a pain score greater than or equal to 4 on a 0-10 numerical pain scale
* Subjects must be willing and able to complete safety and efficacy diaries.
* An escort must be available to pick up the subject at the end of at the end of the surgical/dosing visit (Visit #2)
* In the opinion of the investigators or research coordinators, subjects must be willing and able to understand and comply with study procedures, including completing safety and efficacy diaries at home.
* Able and willing to provide written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* Female subjects who are pregnant or nursing a child.
* Subjects who have received an investigational drug or used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening.
* Subjects who are sensitive or allergic to ibuprofen, acetaminophen, or their components.
* Subjects who are sensitive or allergic to aspirin or other NSAIDs.
* Subjects who are sensitive or allergic to oxycodone or other opioids (excluding nausea and constipation).
* Presence of a serious medical condition (e.g. poorly controlled hypertension or diabetes, gastrointestinal disorders such as bleeding ulcer, coagulation or bleeding disorders, significantly impaired cardiac, renal, hepatic, respiratory, or thyroid function) that according to the investigator may interfere with interpretation of the study results or compromise the safety of a potential subject.
* Acute local infection at the time of surgery that could confound post-surgical evaluation.
* Use of any confounding prescription or non-prescription drug within 24 hours of the surgical procedure, including analgesics, sedating antihistamine, sedative, alcohol, or CNS/psychotropic agents (i.e. sleep aids, benzodiazepines, performance/attention enhancers, marijuana, anti-depressants). Hormonal contraceptives, hormone replacement therapy (including males taking testosterone as a hormone replacement to treat a documented low testosterone level), or thyroid replacement hormones are allowed. Individuals taking other/additional chronic stable medications can be considered on a case-by-case basis for inclusion in the study if agreed upon by judgment of the investigator.
* Subjects who have taken NSAIDs, including acetaminophen, or other medications for pain, including aspirin or aspirin-containing products within 1 week of study drug administration.
* Subjects who routinely consume high doses of antioxidant vitamins daily (vitamin C > 1000mg, Vitamin E > 400IU, Beta Carotene > 1000IU, Vitamin A > 5000IU, Selenium > 200mcg, Folic Acid > 1mg) during the 2 weeks prior to the start of the study.
* Subjects with any abnormal laboratory value or physical finding that according to the investigator may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject.
* Subjects who have a history of abuse of narcotics, street drugs, prescription sleeping pills, based upon history and judgment of the Investigator.
* Subjects who are unwilling to provide a blood sample for genetic analyses.
* Employees of the principal investigator, sub-investigators, or relative of an employee who is directly involved in this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Analgesic response | Up to 7 days after third molar extraction
  Use of opioid rescue medication

SECONDARY OUTCOMES:
Ibuprofen plasma concentrations | Up to 7 days
  Assessed by measuring the amount of ibuprofen in plasma
Acetaminophen plasma concentrations | Up to 7 days
  Assessed by measuring the amount of acetaminophen in plasma
Gene expression profiling | Up to 7 days
  mRNA levels will be measured in peripheral blood mononuclear cells
COX-1 activity | Up to 7 days
  COX-1 activity will be measured ex vivo using a whole blood assay and in vivo by quantifying concentrations of prostaglandin metabolites in urine.
COX-2 activity | Up to 7 days
  COX-2 activity will be measured ex vivo using a whole blood assay and in vivo by quantifying concentrations of prostaglandin metabolites in urine.
DNA sequencing | 1 day
  Assessment of genetic variation
Urinary metabolomics | Up to 7 days
  Assessed by measuring levels of metabolites in urine
Plasma metabolomics | Up to 7 days
  Assessed by measuring levels of metabolites in plasma
Composition of the gut microbiome | 1 day
  Assessed by evaluating the microbes present in a stool sample
Composition of the oral microbiome | 1 day
  Assessed by evaluating the microbes present in an oral swab
Pain intensity score | Up to 7 days
  Rating of pain from 0 (no pain) to 10 (worst imaginable pain)
Inflammatory mediator profiling | Up to 7 days
  Assessment of cytokines in plasma
C-reactive protein | Up to 7 days
  Assessment C-reactive protein in serum
Procalcitonin levels | Up to 7 days
  Assessment of procalcitonin in serum
Complete blood count with differential | Up to 7 days
  Assessment of proportions of red blood cells, white blood cells, and platelets in whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Tilo Grosser, MD, Principal Investigator — University of Pennsylvania; Katherine N Theken, PharmD, PhD, Principal Investigator — University of Pennsylvania; Elliot V Hersh, DMD, MS, PhD, Principal Investigator — University of Pennsylvania; John Farrar, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman JW. The prophylactic extraction of third molars: a public health hazard. Am J Public Health. 2007 Sep;97(9):1554-9. doi: 10.2105/AJPH.2006.100271. Epub 2007 Jul 31. PMID 17666691
- [Background] Gauger EM, Gauger EJ, Desai MJ, Lee DH. Opioid Use After Upper Extremity Surgery. J Hand Surg Am. 2018 May;43(5):470-479. doi: 10.1016/j.jhsa.2018.02.026. Epub 2018 Mar 27. PMID 29602656
- [Background] Maughan BC, Hersh EV, Shofer FS, Wanner KJ, Archer E, Carrasco LR, Rhodes KV. Unused opioid analgesics and drug disposal following outpatient dental surgery: A randomized controlled trial. Drug Alcohol Depend. 2016 Nov 1;168:328-334. doi: 10.1016/j.drugalcdep.2016.08.016. Epub 2016 Sep 20. PMID 27663358
- [Background] Thiels CA, Anderson SS, Ubl DS, Hanson KT, Bergquist WJ, Gray RJ, Gazelka HM, Cima RR, Habermann EB. Wide Variation and Overprescription of Opioids After Elective Surgery. Ann Surg. 2017 Oct;266(4):564-573. doi: 10.1097/SLA.0000000000002365. PMID 28697049
- [Background] Substance Abuse and Mental Health Services Administration (US); Office of the Surgeon General (US). Facing Addiction in America: The Surgeon General's Report on Alcohol, Drugs, and Health [Internet]. Washington (DC): US Department of Health and Human Services; 2016 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK424857/ PMID 28252892
- [Background] Compton WM, Jones CM, Baldwin GT. Relationship between Nonmedical Prescription-Opioid Use and Heroin Use. N Engl J Med. 2016 Jan 14;374(2):154-63. doi: 10.1056/NEJMra1508490. No abstract available. PMID 26760086
- [Background] Cooper SA, Engel J, Ladov M, Precheur H, Rosenheck A, Rauch D. Analgesic efficacy of an ibuprofen-codeine combination. Pharmacotherapy. 1982 May-Jun;2(3):162-7. doi: 10.1002/j.1875-9114.1982.tb04528.x. PMID 6763202
- [Background] Hersh EV, Levin LM, Adamson D, Christensen S, Kiersch TA, Noveck R, Watson G 2nd, Lyon JA. Dose-ranging analgesic study of Prosorb diclofenac potassium in postsurgical dental pain. Clin Ther. 2004 Aug;26(8):1215-27. doi: 10.1016/s0149-2918(04)80033-x. PMID 15476903
- [Background] Hersh EV, Levin LM, Cooper SA, Doyle G, Waksman J, Wedell D, Hong D, Secreto SA. Ibuprofen liquigel for oral surgery pain. Clin Ther. 2000 Nov;22(11):1306-18. doi: 10.1016/s0149-2918(00)83027-1. PMID 11117655
- [Background] Desjardins PJ, Black PM, Daniels S, Bird SR, Fitzgerald BJ, Petruschke RA, Tershakovec A, Chang DJ. A randomized controlled study comparing rofecoxib, diclofenac sodium, and placebo in post-bunionectomy pain. Curr Med Res Opin. 2004 Oct;20(10):1523-37. doi: 10.1185/030079904X3069. PMID 15462686